CLINICAL TRIAL: NCT04867993
Title: Amikacin Pharmacokinetics to Optimize Dosing Recommendations and Patho(Physiological) Considerations in Neonates With Perinatal Asphyxia Treated With Hypothermia
Brief Title: Amikacin Pharmacokinetics to Optimize Dosing Recommendations in Neonates With Perinatal Asphyxia Treated With Hypothermia
Acronym: Amicool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sarajevo (Other)
Collaborators: KU Leuven (Other); Amsterdam UMC, location VUmc (Other); Leiden University Medical Center (Other); University Clinical Center Tuzla (Other)
Responsible Party: Principal Investigator, Sabina Terzic, MD PhD, Assistant professor, University of Sarajevo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0901-2-864/18
Record Dates: First submitted 2021-02-24; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Asphyxia Neonatorum
Keywords: Amikacin; Pharmacokinetics; Hypothermia; Newborn
MeSH Terms: conditions — Asphyxia Neonatorum; Hypothermia | interventions — Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- asphyxiated neonates treated with amikacin and hypothermia (Active Comparator): Amikacin (Likacin®; 500 mg/2mL vial; Lisapharma S.p.A., Erba, Italy) is given to the neonate, as an IV infusion via umbilical vein over 20 min by use of a syringe-pump (Braun; B. Braun Medical Inc., Bethlehem, PA USA). Infusion is followed by slow 0.5 mL Sodium chloride 0.9% flush.
  Interventions: Drug: Amikacin
- asphyxiated neonates treated with amikacin (Placebo Comparator): Amikacin (Likacin®; 500m g/2mL vial; Lisapharma S.p.A., Erba, Italy) is given to the neonate, as an IV infusion via umbilical vein over 20 min by use of a syringe-pump (Braun; B. Braun Medical Inc., Bethlehem, PA USA). Infusion is followed by slow 0.5 mL Sodium chloride 0.9% flush.
  Interventions: Drug: Amikacin

INTERVENTIONS:
Drug: Amikacin — 15 mg/kg/36h

SUMMARY:
As a part of a project on perinatal clinical pharmacology, the primary aim of the present project is to study amikacin pharmacokinetics (PK) and physiology in asphyxiated neonates treated with therapeutic hypothermia and to provide amikacin dosing recommendations, which will be validated prospectively. For this purpose, we aim to first collect retrospective data on amikacin available in neonates treated with hypothermia in the neonatal intensive care unit (NICU)s in Leuven and Amsterdam, and consequently to propose the dosing regimen to be used in the prospective amikacin PK study at our NICU in University Clinical Center (UCC) Sarajevo. At our NICU we aim to collect amikacin PK observations and other covariates in at least 40 neonates while treated with hypothermia and after re-warming period (a paired analysis), and in asphyxiated neonates not treated with hypothermia (control group).

We hereby will use a stepwise approach, as initially used to develop and to validate an amikacin dosing regimen in preterm and term neonates (De Cock RFW et al., 2012, Smits A et al, 2015).

A 3-step approach will be used, of which different parts will be conducted in different contributing hospitals:

1. Retrospective evaluation of amikacin therapeutic drug monitoring (TDM) in asphyxiated neonates treated with hypothermia (University hospital Leuven, VUmc Amsterdam)
2. Development of population PK model derived amikacin dosing recommendation
3. Prospective PK study with validation of the new dosing regimen (UCC Sarajevo, UCC Tuzla)

DETAILED DESCRIPTION:
Step 1: Retrospective evaluation of amikacin TDM in asphyxiated neonates treated with hypothermia (University hospital Leuven, VUmc Amsterdam)

1.1 Study patients All neonates admitted to the NICUs of the VUmc Amsterdam and University hospital Leuven who underwent treatment with hypothermia for perinatal asphyxia and who received amikacin during routine care were considered for inclusion in this retrospective analysis if TDM observations were available. Patients hospitalized between January 2010 and December 2015 were eligible for inclusion. Neonates already included in the Pharmacool trial (de Haan et al BMC Pediatrics 2012), were excluded.

Clinical characteristics at birth [gestational age (GA, weeks), birth bodyweight (grams), Apgar score at 1, 5 and 10 minutes after birth, as well as characteristics at the moment of amikacin TDM [postmenstrual age (PMA, weeks), postnatal age (PNA, days), current bodyweight (grams), concurrent ibuprofen (yes/no) or inotropic drugs (yes/no), respiratory support (i.e. continuous positive airway pressure or mechanical ventilation, yes/no), mechanical ventilation (conventional or high-frequency, yes/no) were retrospectively extracted from the patient files. Additionally, blood culture results at the start of amikacin therapy were collected from the individual laboratory reports. The daily nursing progress reports were used to collect amikacin prescription (dose and interval) data.

1.2 Amikacin dosing regimen

* University hospital Leuven: Up to July 2011, amikacin dosing was based on Langendries JP et al, 1998. Since July 2011, the simplified model-based dosing regimen published by De Cock RFM et al, 2012) was used. Since July 2014, an adapted dosing regimen based on prospective validation is applied (Smits A et al, 2015). In both regimens, the dosing interval was prolonged with 10 hours when ibuprofen was co-administered or when asphyxia was diagnosed/considered by the treating physician.
* Vumc Amsterdam: Up to 24 March 2015 amikacin dosing was 12 mg/kg/dose. Interval (24 hours or 36 hours) was determined based on TDM value and subsequent clearance calculation (see below). From 24 March 2015 amikacin dosing was 15 mg/kg/dose.

1.3 Drug administration and TDM sampling

* University hospital Leuven: amikacine (Bristol-Myers Squibb) is administered intravenously over 20 minutes. As part of routine clinical care, blood samples for amikacin TDM are collected just before (trough) administration of the second dose. In a case of unexpected results or after dosing adaptation, additional TDM samples are collected, based on the decision of the treating physician.
* Vumc: Amikacine (Bristol-Meyers Squib, and recently amikacine Hospira) is administered intravenously over 60 minutes. As part of routine clinical care, the first amikacin TDM sample is taken at least 6 h - but preferably 12-18 h - after the first amikacin administration. This blood sampling is preferably performed during fixed moments at the neonatal department. Based on the amikacin dosing and TDM plasma concentration of the patient, a dosing adaptation is suggested by the pharmacy department, according to the maximum a posteriori Bayesian fitting method, using the MW/Pharm computer program version 3.6 (Mediware, Groningen, the Netherlands). This approach allows variability in TDM sampling time, between and within patients. The predicted target trough level is < 5 mg/L (http://tdm-monografie.org/monografie/amikacine).

1.4 Amikacin assay

* University hospital Leuven: Until 31 May 2012, amikacin concentrations were measured with fluorescence polarization immunoassay (Abbott TDx kit, Abbott Laboratories, Diagnostics Division, Abbott Park, IL, USA). The lower limit of quantification (LLOQ) was 0.8 mg/L. The coefficient of variation (CV) was < 5% (assessed at 5, 15, and 30mg/L). From 31 May 2012, amikacin quantification was based on a kinetic interaction of microparticles in solution (KIMS) immunoassay (Roche/Hitachi Cobas c systems, Roche Diagnostics GmbH, Mannheim, Germany). Also in this essay, the LLOQ was 0.8 mg/L. The CV was < 4%.
* Vumc: Until September 2011, amikacin plasma concentrations were measured with fluorescence polarization immunoassay (Abbott TDx-FLx, Abbott Diagnostics, Abbott Park, IL, USA). The LLOQ was 0.8 mg/L. The CV was < 5% (assessed at 5, 15 and 30m g/L). From September 2011, amikacin quantification was based on a particle-enhanced turbidimetric inhibition immunoassay (PETINIA) (ARCHITECT cSystems, Abbott, Abbott Laboratories Inc, Abbott Park, IL, USA). The limit of quantification for this amikacin assay was 2.0 µg/mL. The coefficient of variation was < 4%.

1.5 Pharmacokinetic analysis The retrospectively collected amikacin TDM values of University hospital Leuven and VUmc Amsterdam will be added to a previously collected dataset of (near)term neonates receiving amikacin but not underwent hypothermia treatment (Smits A et al, 2015). All data will be implemented in the previously developed amikacin population PK model (De Cock R et al, 2012).

Step 2: Development of population PK model derived amikacin dosing recommendation Since a relevant number of neonates treated with hypothermia will be included, we hereby aim to compare pharmacokinetic parameters (clearance, CL, volume of distribution, Vd) of this subgroup of neonates with those of term cases not treated with hypothermia (Smits A et al, 2015). Subsequently, we aim to derive an appropriate model-based dosing regimen to be considered during hypothermia in (near) term cases.

Step 3. Prospective PK study with validation of the new dosing regimen (UCC Sarajevo and UCC Tuzla)

A prospective observational cohort study conducted in NICU with the following aims:

Primary aims:

* to collect amikacin PK observations, renal elimination characteristics and other covariates in at least 40 asphyxiated neonates while treated with hypothermia and after the re-warming period (a paired analysis) (UCC Sarajevo) and in 40 asphyxiated neonates treated with amikacin but not treated with hypothermia (control group, UCC Tuzla)
* validation of the new dosing regimen

Secondary aims of this prospective study are:

* to evaluate amikacin pharmacodynamics (PD) characteristics (minimal inhibitory concentration, MIC90)
* to document the adverse effects of hypothermia (UCC Sarajevo)

3.1 Study patients Asphyxiated neonates routinely treated with IV amikacin and therapeutic hypothermia (NICU UCC Sarajevo) and asphyxiated neonates treated with IV amikacin but not treated with hypothermia (control group, NICU UCC Tuzla) will be included in the study after parental informed written consent is obtained.

3.2 Amikacin dosing regimen

The amikacin dosing regimen that is routinely used in our unit is based on NeoFax® (2009 version) and depends on PMA as follows:

• PMA of equal or more than 35 weeks, 15 mg/kg/24 h with an additional dosing interval increase of 6 h for all ages if ibuprofen was co-administered or in the setting of perinatal asphyxia The dosing regimen (current dosing interval +12 h, 15 mg/kg/36h) derived from asphyxiated neonates treated with hypothermia in Leuven and Amsterdam (step 1-2) will be used in the prospective part of this study (step 3).

3.3 Drug administration and blood sampling Amikacin (Likacin®; 500 mg/2mL vial; Lisapharma S.p.A., Erba, Italy) is given to the neonate, as an IV infusion via umbilical vein over 20 min by use of a syringe-pump (Braun; B. Braun Medical Inc., Bethlehem, PA USA). Infusion is followed by slow 0.5 mL Sodium chloride 0.9% flush.

The collection of samples will be obtained to the current clinical and nursing standard procedures at both NICUs. Blood samples for amikacin TDM and corresponding creatinine concentrations will be collected by venous line via umbilical catheter while collecting the sample for other laboratory findings according to the protocol, 6 minutes before ("trough", the Ctrough) the second, third, fourth and fifth dose of amikacin, than 1h after the initiation of administration ("near peak", the maximal concentration, Cmax) of the second, third and fourth dose of amikacin, approximately 40 min after the 20-min IV infusion (Allegaert K, 2004; Langhendries JP, 1998).

Blood samples (<0.5 mL) will be collected in heparinized tubes. The recommendations for the maximum predefined total amount of blood available for research purposes in a single neonate is 1.0 mL/kg and will be respected.

Blood samples will be centrifuged immediately after collection and subsequently stored at -80°C until analysis. Paired amikacin and creatinine concentrations will be determined.

3.5 Amikacin and creatinine assays Amikacin serum will be determined based on a particle-enhanced turbidimetric inhibition immunoassay (PETINIA) (ARCHITECT cSystems, Abbott, Abbott Laboratories Inc, Abbott Park, IL, USA).

Plasma/serum creatinin concentration will be quantified either by using the "Jaffa method" in Sarajevo or by using the "corrected Jaffa method" in Tuzla.

MIC90 for amikacin will be determined in each Sarajevo and Tuzla NICU before the dosing.

3.6 Pharmacokinetic analysis A compartmental pharmacokinetics approach will be performed at the Department of Pharmacology, Clinical Pharmacology and Toxicology, Medical faculty, University of Sarajevo, B&H.

The population pharmacokinetics approach, comparing the data on PK already reported in neonates will be performed at Leiden Academic Centre for drug research, Leiden University, The Netherlands.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for hypothermia group (University Clinical Centre Sarajevo)

* signed parental informed written consent
* newborn with GA ≥36 weeks
* newborn to whom amikacin is administered by intravenous route for clinical indications
* newborn with perinatal asphyxia treated with hypothermia

Inclusion criteria for control group (University Clinical Centre Tuzla)

* signed parental informed written consent
* newborn to whom amikacin is administered by intravenous route for clinical indications
* newborn with GA ≥36 weeks
* newborn with perinatal asphyxia defined following Bristol hypothermia protocol from 2015

  * Apgar score of ≤5 at 10 minutes after birth OR
  * Continued need for resuscitation, including endotracheal or mask ventilation, at 10 min after birth OR
  * Acidosis defined as either umbilical cord pH or any arterial, venous or capillary pH within 60 min of birth pH<7.00 OR
  * Base deficit ≥-16 mmol/L in umbilical cord blood sample or any blood sample within 60 minutes of birth (arterial or venous blood)

Non-inclusion criteria for both groups

* no parental informed consent
* the presence of congenital hepatic or renal pathology
* no central venous or arterial line in situ for non-invasive blood sampling procedures

Exclusion criteria for both groups

* parental informed consent withdrawal
* the occurrence of clinical reasons to stop blood sampling

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 5 years
  the first plasma concentration measured after the dosing
Minimum Plasma concentration (Ctrough) | 5 years
  the last plasma concentration measured after the dosing
Area under the plasma concentration versus time curve (AUC) | 5 years
  Area under the plasma concentration versus time curve calculated based on a trapezoidal rule
Clearance (CL) | 5 years
  Clearance of the drug, seen from the last part of the concentration-time curve
Volume of distribution (Vd) | 5 years
  Volume of distribution of the drug, seen from the early part of the concentration-time curve
Minumum inhibitory concentration (MIC 90) | 5 years
  concentration of the drug needed to inhibit the growth of 90% of isolates
Creatinine clearance | 5 years
  clearance of the creatinine calculated by different formulas

SECONDARY OUTCOMES:
adverse effects of hypothermia | 5 years
  adverse outcomes of hypothermia

CONTACTS AND LOCATIONS:
Overall Officials: Karel Allegaert, MD PhD, Study Chair — Catholic University Leuven, Belgium
Locations (1):
- Pediatric Clinic, University Clinical Centre Sarajevo, Sarajevo, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Cock RF, Allegaert K, Schreuder MF, Sherwin CM, de Hoog M, van den Anker JN, Danhof M, Knibbe CA. Maturation of the glomerular filtration rate in neonates, as reflected by amikacin clearance. Clin Pharmacokinet. 2012 Feb 1;51(2):105-17. doi: 10.2165/11595640-000000000-00000. PMID 22229883
- [Background] Smits A, De Cock RF, Allegaert K, Vanhaesebrouck S, Danhof M, Knibbe CA. Prospective Evaluation of a Model-Based Dosing Regimen for Amikacin in Preterm and Term Neonates in Clinical Practice. Antimicrob Agents Chemother. 2015 Oct;59(10):6344-51. doi: 10.1128/AAC.01157-15. Epub 2015 Jul 27. PMID 26248375
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22229883-maturation-of-the-glomerular-filtration-rate-in-neonates-as-reflected-by-amikacin-clearance/?from_single_result=De+Cock+RFW%2C+Allegaert+K%2C+Schreuder+MF.%2C+Sherwin+CM%2C+de+Hoog+M%2C+van+den+Anker+JN.%2C+Danhof+Mand+Knibbe+CAJ.+Maturation+of+the+Glomerular+Filtration+Rate+in+Neonates%2C+as+Reflected+by+Amikacin+Clearance.+Clin+Pharmacokinet.+2012%3B+51%282%29%3A105-17.+doi%3A+10.2165%2F11595640-000000000-00000.
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26248375-prospective-evaluation-of-a-model-based-dosing-regimen-for-amikacin-in-preterm-and-term-neonates-in-clinical-practice/?from_single_result=Smits+A%2C+De+Cock+RF%2C+Allegaert+K%2C+Vanhaesebrouck+S%2C+Danhof+M%2C+Knibbe+CA.+Prospective+Evaluation+of+a+Model+Based+Dosing+Regimen+for+Amikacin+in+Preterm+and+Term+Neonates+in+Clinical+Practice.+Antimicrob+Agents+Chemother.+2015%3B+59%2810%29%3A6344-51.